CLINICAL TRIAL: NCT02871973
Title: Sit Down and Play: A Primary Care-Based Program to Promote Positive Parenting Practices
Brief Title: Primary Care-based Program to Enhance Positive Parenting Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Reshma Shah, MD, Assistant Professor of Clinical Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2014-0337_1; UL1TR000050 (NIH)
Record Dates: First submitted 2016-08-10; First posted 2016-08-18 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Parenting; Development; Language; Children
Keywords: parenting; child development; language
MeSH Terms: conditions — Language

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SDP (Experimental): Families randomized to intervention group will receive Sit Down and Play while they wait in the waiting room to be seen by their primary care provider at current and subsequent well-child visit.
  Interventions: Behavioral: Sit Down and Play
- CDC Handout (Active Comparator): Families in the control group will receive the Center for Disease Control and Prevention (CDC) Handout at enrollment.
  Interventions: Behavioral: Handout

INTERVENTIONS:
Behavioral: Sit Down and Play — Sit Down and Play (SDP) is designed to be a brief, low-cost intervention that incorporates key theoretical constructs to elicit positive parenting behaviors. It is intended to be delivered by existing clinical staff, nonprofessionals, or volunteers during each of the eight well-child visits between 2-24 months of age while a family waits to be seen by their pediatrician in the examination room.
  Arms: SDP
Behavioral: Handout — Handouts developed by Center for Disease Control and Prevention (CDC) to provide information regarding age-specific early childhood milestones
  Arms: CDC Handout

SUMMARY:
The objective of this research is to conduct a small randomized pilot study to evaluate the feasibility of Sit Down and Play (SDP), a brief, low-cost program delivered in the primary care setting to enhance parent-child interactions and explore potential impacts on parenting behaviors.

DETAILED DESCRIPTION:
Enriching parenting behaviors in early childhood promotes child development and offers a promising strategy to reduce future educational disparities. However, current interventions are limited by cost and have not been widely disseminated. Recognized as a target for research to improve early childhood development and school readiness among at-risk families, the primary care setting offers an ideal opportunity to reach the millions of children living in poverty.However, what remains unknown is how to more efficiently leverage the primary care setting to deliver a sustainable and effective preventive intervention to promote positive parenting behaviors and encourage early childhood development in low-income families. Therefore, the investigators designed Sit Down and Play (SDP) a brief parent-directed program delivered in the primary care setting. Modeled after the widely disseminated literacy program Reach Out and Read and grounded in social cognitive theory, SDP is intended to take place during each pediatric well-child visit occurring in a child's first two years with the goal of promoting positive parenting behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Parent is 18 years or older
* Child is present for a 2, 4, or 6 month well-child visit
* Adult present with child at appointment is parent/caregiver of child

Exclusion Criteria:

* Parent is non-English speaking
* Child is acutely sick

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Caregiver's participation in cognitively stimulating activities such as reading and playing using self-report measure StimQ | 3-4 months post-enrollment
Parental Self-Efficacy as measured by Parenting Sense of Competence Scale | 3-4 months post-enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Reshma Shah, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shah R, Kennedy S, Clark MD, Bauer SC, Schwartz A. Primary Care-Based Interventions to Promote Positive Parenting Behaviors: A Meta-analysis. Pediatrics. 2016 May;137(5):e20153393. doi: 10.1542/peds.2015-3393. Epub 2016 Apr 19. PMID 27244800
- [Background] Shah R, Sobotka SA, Chen YF, Msall ME. Positive Parenting Practices, Health Disparities, and Developmental Progress. Pediatrics. 2015 Aug;136(2):318-26. doi: 10.1542/peds.2014-3390. PMID 26216325